CLINICAL TRIAL: NCT04022057
Title: The Impact of a Preoperative Nerve Block in Foot and Ankle Surgery on the Consumption of Sevoflurane
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00092857
Record Dates: First submitted 2019-07-08; First posted 2019-07-16 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Ankle Arthropathy; Anesthesia; Functional; Ankle Arthritis
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized controlled, prospective
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-GA (Active Comparator): 10 mL of 1% ropivacaine injection before the start of surgery and 10 ml of 5% dextrose injection at the end of surgery through both the popliteal and the saphenous catheter
  Interventions: Drug: Ropivacaine injection; Drug: Dextrose 5
- Post-GA (Sham Comparator): 10 mL of 5% dextrose injection before the start of surgery and 10 ml of 1% ropivacaine injection at the end of surgery through both the popliteal and the saphenous catheter
  Interventions: Drug: Ropivacaine injection; Drug: Dextrose 5

INTERVENTIONS:
Drug: Ropivacaine injection — Local anesthetic injection
Drug: Dextrose 5 — Sham Injection

SUMMARY:
Reconstructive foot and ankle surgery is performed under general anesthesia. Included in this spectrum of surgery are ankle arthroplasties, various fusions, corrective arthrodesis, and more. Pain control for after the surgery can be achieved purely with intravenous and oral pain medication or in combination with freezing of the nerves. Nerve freezing (nerve block) placed before surgery has the potential to substantially reduce the amount of inhaled anesthetic given to the patient during surgery. This can benefit the patient with being more awake and crisp more quickly after surgery. It can also reduce cost to the system. A further benefit which has received very little attention so far, is that reducing the amount of inhaled anesthetic given also lowers the environmental footprint created by the anesthetic. For the region of the foot and ankle to be fully frozen, both the sciatic nerve and the saphenous nerve must be successfully blocked. Sciatic nerve blockade is most commonly achieved by blocking the nerve in the popliteal fossa. This block is named popliteal nerve block.

The investigators will examine and quantify the amount of inhaled anesthetic used for each case and will compare how the consumption is affected by whether the nerve blocks are applied before or after surgery. Patients will have two nerve block catheters (popliteal and saphenous catheter) placed under ultrasound-guidance prior to the case by an experienced and specifically trained anesthesiologist. The catheters will be loaded with a solution to which the anesthesiologist is blinded. It will either be local anesthetic or 5% dextrose (sham). The general anesthetic will be conducted according to a research protocol with anesthetic depth being the targeted endpoint. Measurements of the required MAC-Value (minimum alveolar concentration) of inhaled anesthetic will be recorded every five minutes by a study team member. At the end of the case the anesthesiologist will be unblinded to the solution. Should the patient have received sham initially, they will now receive the full dose of local anesthetic prior to being woken up.

DETAILED DESCRIPTION:
Following ethics approval, eligible patients meeting the inclusion/exclusion criteria will be consented in pre-assessment unit or day surgery at least 2 hours prior to surgery. Patients will then be randomized into two groups:

1. Popliteal and saphenous nerve block catheter insertion with 10 mL 1% ropivacaine injection into each (Treatment group)
2. Popliteal and saphenous nerve block catheter insertion with 10 mL 5% dextrose injection into each (Sham)

All syringes will be blinded to the anesthesiologist in the case. Each patient will have two syringes for before and for after surgery - one set for treatment and one sham. Depending on the randomization they will get first one before surgery and then the other after surgery. Popliteal and saphenous nerve block catheters will be inserted under ultrasound guidance using the catheter-over-needle technique whereby the location of the tip of the catheter can be easily determined. All nerve block catheters will be performed by experienced acute pain physicians who have been performing interscalene blocks under ultrasound guidance for at least 5 years. Successful catheter placement will be verified by following the spread of the injectate, which will occur just before induction of general anesthesia in the operating room. Induction of general anesthesia will follow a standardized protocol with the intravenous administration of sufentanil 0.2 mcg/kg, propofol 2 mg/kg, and rocuronium 0.5 mg/kg. General anesthesia will be maintained with sevoflurane, which will be age-adjusted to 1.0 minimum alveolar concentration (MAC) to begin the case and then adjusted from there as per protocol. Sedline, Masimo® will be used to monitor the depth of anesthesia. The intraoperative patient state index (PSI) target will be 25 - 50. As per protocol, adjustments of the age-adjusted MAC will be performed as follows at every measuring point:

A PSI of either below 25 or of over 50 will always be treated with an adjustment of the age-adjusted MAC value. The same is done if the heart rate and/or the blood pressure is outside of +/- 20% of baseline. The primary goal is to treat any of the above changes with an adjustment to the age-adjusted MAC value. The anesthesiologist will always be able to administer an analgesic, should this be clinically necessary. The patient will be given a bolus of 1 mcg/kg of remifentanil and this will be recorded. The age-adjusted MAC value will be recorded every 5 minutes until the anesthesiologist reduces the anesthetic in preparation for extubation. At the conclusion of surgery and before general anesthesia is ended, the patients will receive the second set of solutions injected into their catheters.

Postoperatively, patients will go to post-anesthesia care unit (PACU). The distribution of the sensory or motor block will then be checked and recorded 30 minutes after arriving in PACU in both groups. The numerical rating scale (NRS) for pain will also be recorded in PACU at 0, 15, 30 and 45 minutes. The patients will there be assessed by members of the acute pain service team and treated as necessary before being transferred to the ward.

The patient, operating room anesthesiologist and the data collection personnel will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective reconstructive foot and ankle surgery
* Patients eligible for popliteal and saphenous nerve block
* All adults 18 years of age or older
* Capable to give consent

Exclusion Criteria:

* Patients who are unable to give consent
* Local anaesthetic allergy
* Hemidiaphragm paresis on the contralateral side to the block/surgery site
* Bleeding diathesis
* Coagulopathy
* Pre-existing neurological deficits
* Patients with a Body Mass Index >35
* Patients with significant comorbidities, physiological limitations, and allergies that are unable to tolerate the protocolized induction and maintenance of anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All gender identification and self-representation is accepted
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Age-adjusted MAC of sevoflurane per hour | Intraoperative measurement done at the end of anesthetic
  The average age-adjusted end- tidal minimum alveolar concentration (MAC) will be calculated by averaging the end tidal MAC required to maintain the depth of anesthesia as measured by PSI between 25-50 intra-operatively. This will be compared between the two groups.

SECONDARY OUTCOMES:
Intraoperative heart rate | Intraoperative period
  Intraoperative heart rate (in beats/minute) will be documented at 5 minute interval and compared between the two groups
Intraoperative opioid use | Intraoperative period
  Intraoperative use of short acting opioid (in microgram/Kg) as per the study protocol will be recorded and compared between the two groups
Postoperative opioid use in PACU | Up to 24 postoperative hours
  Total amount of opioids (in mg of morphine equivalents) in the PACU and over the first 24 postoperative hours will be recorded and compared between the two groups
Maximum pain scores in the first 24 post-operative hours | Up to 24 postoperative hours
  Maximum pain scores will be recorded using numerical rating scale (NRS) of 0-10 (where 0=no pain and 10= maximum pain) on arrival to PACU and at 0,15,30, 45 minutes and at 24 postoperative hours and compared between the two groups
Nausea and vomiting in the first 24 post-operative hours | Up to 24 postoperative hours
  Nausea scores (on a Likert scale of 1-4 where 1 = no nausea, 2= mild nausea, 3= moderate nausea and 4= severe nausea/vomiting will be recorded on arrival to PACU and at 0,15,30, 45 minutes and at 24 postoperative hours and will be compared between the two groups
24 hour opioid consumption | Up to 24 postoperative hours
  Total consumption of opioids (in morphine equivalents) over the first 24 postoperative hours will be recorded and compared between the two groups
The sedation score in PACU | 1st postoperative hour
  Sedation scores will be recorded at 15 minute intervals based on Ramsay sedation scale (1-6) and will be compared between the two groups
Sensory testing of nerves in the distribution of the nerve block ("Cold test") | 1st postoperative hour
  Sensory testing of the L2-S4 dermatomes will be performed in the PACU at 30 minutes of arrival to PACU to document the success of the block
Intraoperative vasopressor usage | Intraoperative period
  Amount and frequency of the intraoperative usage of vasopressor (phenylephrine in micrograms) will be documented and compared between the two groups
Intraoperative Mean blood pressure | Intraoperative period
  Intraoperative mean blood pressure (in mm Hg) will be documented at 5 minute interval and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Vivian HY Ip, MD, Study Director — University of Alberta; Lora Pencheva, MD, Study Director — University of Alberta; Rakesh V Sondekoppam, MD, Study Chair — University of Alberta; Timur JP Özelsel, MD, DESA, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada